CLINICAL TRIAL: NCT00383864
Title: Randomized Study on the Efficacy and Safety of Pegylated Interferon and Ribavirin in Hepatitis C Virus Infection After Liver Transplantation
Brief Title: Pegylated Interferon and Ribavirin in Hepatitis C Virus Infection After Liver Transplantation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEG/RBV POST-TOH
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Hepatitis C
Keywords: liver fibrosis; portal pressure; antiviral therapy
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis | interventions — Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon and ribavirin

SUMMARY:
The purpose of this study was to evaluate the efficacy (and safety) of antiviral therapy in patients with chronic hepatitis C after liver transplantation. The only approved drugs for treatment of hepatitis C are pegylated interferon and ribavirin.

DETAILED DESCRIPTION:
Hepatitis C recurrence after liver transplantation remains the main cause of graft loss after liver transplantation. Several strategies can be used to prevent or treat hepatitis C in the setting of liver transplantation. There are no controlled studies evaluating the efficacy and safety of antiviral treatment (using pegylated interferon and ribavirin) in liver transplant recipients. The main endpoint of this study was: 1) histological outcomes (effect of antiviral treatment on disease progression, i.e. liver fibrosis). The secondary endpoint were 1) Sustained virological response (persistent HCV-RNA clearance) and 2) Safety of pegylated interferon and ribavirin

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C defined by liver biopsy and presence of HCV-RNA
* More than 6 months from liver transplantation
* Written inform consent

Exclusion Criteria:

* Severe hepatitis C recurrence (F3-F4 fibrosis stage, cholestatic hepatitis)
* Double liver-kidney transplantation
* Leucopenia (2000) or thrombocytopenia (40.000)
* Anemia (Hemoglobin lower than 10 g/dL)
* Renal failure (creatinine > 2 mg/dL)
* Autoimmune disease
* All contraindications for interferon and ribavirin therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2001-07; Study Completion 2006-03

PRIMARY OUTCOMES:
Histological improvement (decrease in at least one fibrosis stage in follow-up liver biop

SECONDARY OUTCOMES:
Sustained virological response (persistent HCV-RNA negativation)
Safety of antiviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Forns, MD, Principal Investigator — Liver Unit, Hospital Clinic, Barcelona
Locations (1):
- Liver Unit, Hospital Clinic, Barcelona, Spain

REFERENCES:
- [Derived] Carrion JA, Navasa M, Garcia-Retortillo M, Garcia-Pagan JC, Crespo G, Bruguera M, Bosch J, Forns X. Efficacy of antiviral therapy on hepatitis C recurrence after liver transplantation: a randomized controlled study. Gastroenterology. 2007 May;132(5):1746-56. doi: 10.1053/j.gastro.2007.03.041. Epub 2007 Mar 24. PMID 17484872